CLINICAL TRIAL: NCT05177809
Title: RFC1 Natural History Study
Acronym: RFC1-NHS
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Matthis Synofzik (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Matthis Synofzik, Principal Investigator, Leading Consultant, University Hospital Tuebingen
Organization: University Hospital Tuebingen (Other)
Other Study IDs: RFC1-NHS
Record Dates: First submitted 2021-12-14; First posted 2022-01-05 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Ataxia
Keywords: RFC1; CANVAS; Natural History Study; Biomarker
MeSH Terms: conditions — Ataxia | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — optional biosample collection including blood (DNA, serum, plasma, RNA, PBMC), urine, CSF, skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RFC1: Participants with genetically confirmed RFC1 repeat expansion disease (ORPHA: 504476; OMIM 102579) will be recruited. Target sample size for the RFC1 cohort is 100 participants.
  Interventions: Other: Clinical rating scale to measure ataxia disease severity and progression
- Unrelated healthy controls: Unrelated healthy controls Healthy controls may undergo the same study procedures as the RFC1 cohort. Target sample size for the control cohort is 50.

INTERVENTIONS:
Other: Clinical rating scale to measure ataxia disease severity and progression — SARA is a clinical scale developed by Schmitz-Hübsch et al which assesses a range of different impairments in cerebellar ataxia. The scale is made up of 8 items related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test.
  Other Names: Scale for the Assessment and rating of Ataxia (SARA)
  Groups: RFC1

SUMMARY:
This international, multi-center, multi-modal and prospective observational study aims to determine the phenotypic spectrum and the natural progression of the RFC1 repeat expansion disease, and to seek and validate digital, imaging, and molecular biomarkers that aid in diagnosis and serve as outcome measures in future clinical trials of this novel, but frequent ataxia with late adult-onset.

DETAILED DESCRIPTION:
The investigators will perform an international, multi-center, multi-modal, and registry-based standardized prospective Natural History Study (NHS) in RFC1 repeat expansion disease. Participants will be assessed annually. Study visits with a standardized clinical examination will apply several clinical rating scales, and data will be entered into a clinical database (ARCA Registry; www.ARCA-registry.org) customized to the requirements of this specific study. At all study visits, patients will be asked to donate biosamples; biomaterial collection is optional, and participants can elect to participate in sampling of blood, urine, CSF, and/or a skin biopsy.

Optionally, and depending on local availability at each participating site, additional examinations may be performed including imaging, quantitative movement and speech analysis, vestibular testing, a neuropsychological examination, or examination of swallowing function, all to fully capture the multisystemic presentation of the RFC1 repeat expansion disease.

This study will delineate variable phenotypes of this relatively novel disease, and systematically characterize the longitudinal progression of multi-model biomarkers to determine the most sensitive, comprehensive, and reliable outcomes measures for future therapeutic trials. Here, longitudinal validation of targeted fluid biomarker candidates will be an important part. The multi-modal longitudinal design of the study and its comprehensive assessment will also provide mechanistic insights into the multisystemic evolution of the disease, which will especially allow to track and understand selective as well as overlapping dysfunction of the cerebellum, sensory peripheral nerves, the vestibular system, and additional systems known to be involved in RFC1 disease or 'CANVAS' as its related syndrome.

ELIGIBILITY:
Inclusion Criteria:

* RFC1: genetic diagnosis of bi-allelic pathogenic repeat expansions in RFC1
* Unrelated healthy controls: no signs or history of neurological or psychiatric disease AND
* Written informed consent AND
* Participants are willing and able to comply with study procedures

Exclusion Criteria:

* RFC1: Missing informed consent
* Controls: evidence of neuropathy, neurodegenerative disease, or movement disorder; inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study enrolls probands with clinically manifest and genetically confirmed RFC1 repeat expansion disease, as well as healthy unrelated controls to contrast unspecific, age- or sex-related findings to disease-related specific findings.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of Scale for the Assessment and Rating of Ataxia (SARA) from baseline to 2-year follow-up. | 24 months
  Severity of ataxia in the RFC1 cohort will be assessed by application of the Scale for the Assessment and Rating of Ataxia (SARA). The total score is calculated as the sum of 8 items, yielding a total score between 0 and 40. Hereby, higher SARA scores indicate more severe disease.

SECONDARY OUTCOMES:
Friedreich Ataxia Rating Scale - Activities of Daily Living (FARS-ADL) from baseline to 2-year follow-up. | 24 months
  Impairment in activities of daily living by ataxia, neuropathy, vestibular impairment or other disease features will be assessed in the RFC1 cohort by application of the Activities of Daily Living part of the Friedreich Ataxia Rating Scale (FARS-ADL). The total score is calculated as the sum of 9 items, yielding a total score between 0 and 36. Hereby, higher FARS-ADL scores indicate more severe functional impairment.
Charcot-Marie-Tooth Examination Score Version 2 (CMTESv2) from baseline to 2-year follow-up. | 24 months
  Severity of neuropathy in the RFC1 cohort will be assessed by application of the Charcot-Marie-Tooth Examination Score Version 2 (CMTESv2). The total score is calculated as the sum of 7 items, yielding a total score between 0 and 28. Hereby, higher CMTESv2 scores indicate more severe neuropathy.
Nine-Hole Peg Test (9HPT) from baseline to 2-year follow-up. | 24 months
  Upper limb function in the RFC1 cohort will be quantified by application of the Nine-Hole Peg Test (9HPT). This performance measure yields the mean duration of 2 trials to complete the task with the dominant and non-dominant hand, respectively, with an upper limit of 5 minutes (300 seconds).

OTHER OUTCOMES:
Composite Autonomic Symptom Score (COMPASS-31) at baseline, and eventually from baseline to 2-year follow-up if baseline data supports further use. | 24 months
  Severity of dysautonomia will be assessed by application of the Composite Autonomic Symptom Score (COMPASS-31). The total score is calculated as the weighted sum of 31 questions items, yielding a total autonomic symptom score between 0 and 100. Hereby, higher COMPASS-31 cores indicate more severe dysautonomia. This module is optional in the RFC1 cohort and unrelated healthy controls.
Cerebellar cognitive-affective syndrome scale (CCAS) from baseline to 2-year follow-up. | 24 months
  Severity of cognitive impairment will be assessed by application of the Cerebellar cognitive-affective syndrome scale (CCAS). The total score of 15 items comprises the number of failed items (with 3 or more failed items indicating definite cerebellar cognitive-affective syndrome), and a raw total score between 0 and 120. Hereby, lower CCAS raw cores indicate more severe cognitive impairment. This module is optional in the RFC1 cohort and unrelated healthy controls.
Clinical Assessment of Dysphagia in Neurodegeneration (CADN) from baseline to 2-year follow-up. | 24 months
  Severity of dysphagia will be assessed by application of the Clinical Assessment of Dysphagia in Neurodegeneration (CADN), comprising a history part and an examination with consumption. The total score is calculated as the weighted sum of 11 items, yielding a total score between 0 and 10. Hereby, higher CADN scores indicate more severe dysphagia. This module is optional in the RFC1 cohort.
Video Head Impulse Test (vHIT) from baseline to 2-year follow-up. | 24 months
  Vestibular function will be quantified by application of the Video Head Impulse Test (vHIT) of the horizontal semicircular canals, and eventually the vertical semicircular canals. This test yields the gain (ratio of eye velocity to head velocity) as a measure of vestibular function, yielding total scores between 0 and 1. Hereby, lower gains indicate more severe vestibular impairment. This module is optional in the RFC1 cohort and unrelated healthy controls.
Digital gait and balance assessment from baseline to 2-year follow-up. | 24 months
  Gait and balance will be assessed digitally with body-worn sensors (inertial measurement units), which record acceleration or rotational movements during specific gait and balance tasks. This module is optional in the RFC1 cohort and unrelated healthy controls.
Digital assessment of limb function from baseline to 2-year follow-up. | 24 months
  Motor skills of the upper and lower limb will we assessed digitally with a quantitative motor examination (Q-Motor), which measures contact pressure and position in space during specific motor tasks. This module is optional in the RFC1 cohort and unrelated healthy controls.
Digital Speech Assessment from baseline to 2-year follow-up. | 24 months
  Dysarthria will be assessed using Redenlab audio capture and analysis software. Speakers will complete connected speech, syllable repetition and sustained vowel tasks. Data will be analyzed for measures of voice quality, articulation, breath support, resonance, and prosody. This module is optional in the RFC1 cohort and unrelated healthy controls.
Magnetic resonance imaging (MRI) from baseline to 2-year follow-up. | 24 months
  Structural integrity of the brain and cervical spine will be assessed by application of Magnetic Resonance Imaging (MRI), with a core dataset of T1-weighted, T2-weighted, and diffusion-weighted imaging sequences. This module is optional in the RFC1 cohort and unrelated healthy controls.
Patient-reported outcomes of chronic cough from baseline to 2-year follow-up. | 24 months
  The presence and severity of chronic cough will be assessed with the Cough Severity Visual Analogue Scale and the Leicester Cough Questionnaire as validated patient-reported outcomes and trial endpoints of chronic cough.

CONTACTS AND LOCATIONS:
Overall Officials: Matthis Synofzik, Prof. Dr., Principal Investigator — University Hospital Tübingen; Andreas Traschütz, Dr. Dr., Principal Investigator — University Hospital Tübingen
Locations (10):
- Department of Neuroscience, Central Clinical School, Monash University, Melbourne, Victoria, Australia
- Department of Neurology, Ataxia Unit, Universidade Federal de São Paulo, São Paulo, State of São Paulo, Brazil
- Service de Neurologie, Hôpitaux Universitaires de Strasbourg, Strasbourg, France
- Germany (3):
  - Center for Neurology & Hertie-Institute for Clinical Brain Research, Dept. for Neurodegenerative Diseases, Tübingen, Baden-Wurttemberg
  - German Center for Neurodegenerative Diseases (DZNE), Bonn, North Rhine-Westphalia
  - Department of Neurology University Hospital Schleswig Holstein, Lübeck, Schleswig-Holstein
- Italy (2):
  - Università degli Studi di Napoli 'Federico II', c/o AOU Federico II, Napoli
  - IRCCS Fondazione Stella Maris, Pisa
- Centre of Brain Research Neurogenetics Research Clinic, University of Auckland, Auckland, New Zealand
- Koç University Hospital, KUTTAM-NDAL, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website of the ARCA Registry — http://arca-registry.org